CLINICAL TRIAL: NCT02344251
Title: A Phase II Randomized Trial to Assess the Effectiveness and Safety of the ID-Cap System for Medication Ingestion Monitoring and Enhancing Adherence
Brief Title: Assessing the Effectiveness and Safety of the ID-Cap System for Medication Monitoring and Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO00033472
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Medication Adherence
Keywords: Drug study; Medication compliance
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Other): Adherence measured by MEMS Cap
  Interventions: Device: MEMS Cap
- Group 2 (Other): Adherence measured by ID-Cap technology.
  Interventions: Device: ID-Cap

INTERVENTIONS:
Device: MEMS Cap — MEMS Track Cap records when the medication bottle is opened and closed
  Arms: Group 1
Device: ID-Cap — ID-Cap Tag is an ingestible medical device for detecting the presence of an ingested capsule inside the gastrointestinal (GI) tract.
  Arms: Group 2

SUMMARY:
In pharmacotherapy trials involving drug-dependent individuals, medication compliance is a significant issue, as rates tend to be low and adherence to medication may predict improved outcomes (Baros et al, 2007; McRae et al, 2004; O'Brien et al, 1996; Somoza et al., 2010). However, methods commonly used to determine compliance may result in inaccurate measurement of adherence. In this study, we propose to assess the effectiveness and safety of the ID-Cap System, a novel compliance measurement device, in a healthy population.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to evaluate the acceptability, tolerability, and efficacy of the ID-Cap system in a healthy population. The ID-Cap is an ingestible medical device for detecting the presence of an ingested capsule inside the gastrointestinal (GI) tract.

Participation in the study takes 3 visits over a period of approximately six weeks. The first visit is a screening visit to determine if participants are eligible to participate. After the initial assessment visit, participants will be randomized to one of two groups. Group 1 will have adherence measured by self-report, pill count, and urine riboflavin levels. This group will not receive capsules containing ingestible sensors, but will receive their medication in a bottle capped with a MEMS Track Cap, which records when the medication bottle is opened and closed. Group 2 will receive capsules containing an ingestible sensor and will have adherence measured by self-report, pill count, urine riboflavin levels as needed, and data collected by an ID-Cap reader. Participants randomized to this group will also receive reminder calls and/or text messages to ingest the study medication if a signal is not sent from the ID-Cap reader to the study team within one hour of the scheduled medication administration time. They will also be using biometric identification technology to confirm subject identity, specifically electrocardiogram (ECG).

After the initial screening visit, participants will be required to attend two clinic visits during the six-week study, a randomization visit and a one-week follow-up visit approximately one week after last medication dose.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 and 65 years
* If female and of childbearing potential, must agree to use acceptable methods of birth control for the duration of the trial
* Must consent to random assignment, and be willing to commit to medication ingestion
* Must be able to read and provide informed consent
* Must function at an intellectual level sufficient to allow accurate completion of assessments
* Must have a Body Mass Index (BMI) below 35

Exclusion Criteria:

* Women who are pregnant, nursing, or plan to become pregnant during the course of the study
* Must not have evidence of a significant medical condition which may affect capsule passage through the gastrointestinal tract (including, but not limited to, Crohn's disease, small bowel tumors, intestinal adhesions, ulcerations, and radiation enteritis)
* Must not have a current major psychiatric disorder as these may interfere with assessment measures
* Must not be currently dependent on other substances, with the exception of nicotine or caffeine, within the past 60 days
* Hypersensitivity to riboflavin or any capsule component;
* Individuals with embedded electronic devices
* Patients who, in the investigator's opinion, would be unable to comply with study procedures or assessments, or would be unacceptable study candidates (e.g., poses threat to staff)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee McRae-Clark, PharmD, BCPP, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MEMS Track Cap: Compliance measured by MEMS Cap, riboflavin and self-report.
  MEMS Cap: MEMS Track Cap records when the medication bottle is opened and closed
  Riboflavin: 50 mg
- ID Cap Tag: Compliance measured by riboflavin, self-report, and ID-Cap technology.
  ID-Cap: ID-Cap Tag is an ingestible medical device for detecting the presence of an ingested capsule inside the gastrointestinal (GI) tract.
  Riboflavin: 50 mg
Period: Overall Study
Arm/Group | MEMS Track Cap | ID Cap Tag
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MEMS Track Cap: Compliance measured by MEMS Cap
  MEMS Cap: MEMS Track Cap records when the medication bottle is opened and closed
- ID Cap Tag: Compliance measured by ID-Cap technology
  ID-Cap: ID-Cap Tag is an ingestible medical device for detecting the presence of an ingested capsule inside the gastrointestinal (GI) tract.
- Total: Total of all reporting groups
Arm/Group | MEMS Track Cap | ID Cap Tag | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 11 | 14 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: The primary outcome will be medication adherence as measured by percentage of doses taken among groups.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of doses taken
Groups:
- MEMS Track Cap: Adherence measured by MEMS Cap
  MEMS Cap: MEMS Track Cap records when the medication bottle is opened and closed
- ID Cap: Adherence measured by ID-Cap technology.
  ID-Capsule: ID-Capsule is an ingestible medical device for detecting the presence of an ingested capsule inside the gastrointestinal (GI) tract.
Arm/Group | MEMS Track Cap | ID Cap
Number analyzed (Participants) | 20 | 20
percentage of doses taken | 94.8 [92.2 to 97.3] | 82.8 [76.4 to 89.3]

2. Secondary Outcome: Safety Assessment: Rates of Adverse Events Reported
Description: A secondary outcome will be safety assessment as measured by the percentage of participants reporting adverse events.
Time Frame: 30 days
Measure: Number; unit: percentage of participants reporting AEs
Groups:
- ID Cap: Compliance measured by ID-Cap technology.
  ID-Cap: ID-Cap Tag is an ingestible medical device for detecting the presence of an ingested capsule inside the gastrointestinal (GI) tract.
Arm/Group | MEMS Track Cap | ID Cap
Number analyzed (Participants) | 20 | 20
percentage of participants reporting AEs | 25 | 15

ADVERSE EVENTS:
Time Frame: 4 week medication period
Groups:
- ID Cap Tag: Compliance measured by ID-Cap technology.
  ID-Cap: ID-Cap Tag is an ingestible medical device for detecting the presence of an ingested capsule inside the gastrointestinal (GI) tract.
Arm/Group | MEMS Track Cap | ID Cap Tag
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEMS Track Cap (N=20) | ID Cap Tag (N=20)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) — exact symptom(s) not detailed in AE report
Ringworm (Infections and infestations) | 1 (1) | 0 (0)
Increased urination (Renal and urinary disorders) | 1 (1) | 0 (0)
weight gain (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limited generalizability- participants were primarily MUSC students & staff. The ID Cap system is only available for adherence measurement for solid oral dosage medications. Potential for user error due to the electronic nature of the ID Cap system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT02344251/Prot_SAP_000.pdf